CLINICAL TRIAL: NCT02943122
Title: Prognostic Value of Ambulatory Blood Pressure Monitoring Pattern in Post-Partum Pre-Eclamptic Patients
Brief Title: Ambulatory Blood Pressure Monitoring in Post-Partum Pre-Eclamptic Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: ABPM
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Decrease Maternal Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ambulatory blood pressure monitor

SUMMARY:
Preeclamptic pregnancy is associated with alterations in the left ventricular structure and function and elevation of cardiovascular biomarkers. The alterations are still persistent several months after delivery and are more clearly observed in early-onset and severe Pre-eclampsia

ELIGIBILITY:
Inclusion Criteria:

* All previously healthy women who were diagnosed as preeclampsia.( defined as gestational hypertension ( systolic BP of at least 140 mm Hg and/or a diastolic BP of at least 90 mm Hg on at least two occasions at least 6 hours apart after the 20th week of gestation in women known to be normotensive before pregnancy and before 20 weeks' gestation ) plus proteinuria (300 mg or more per 24-hour period)

Exclusion Criteria:

* Current pregnancy
* Chronic hypertension or any condition requiring the use of antihypertensive medication
* Chronic kidney disease
* Any disease requiring the use of anti-inflammatory medication, diabetes or any other endocrine disease such as hyperthyroidism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: all women suffered from preeclampsia in last pregnancy will be examined 3 months after delivery /or termination
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
number of women with persistent hypertension | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No